CLINICAL TRIAL: NCT06878638
Title: Impact of Intravenous Nitrate Treatment on Antiplatelet Effects of Clopidogrel in Acute Coronary Syndrome Patients: A Pilot Study
Brief Title: Nitrate - Clopidogrel - Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: Bursa Yüksek İhtisas
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Coronary Syndromes
Keywords: Intravenous nitrate; clopidogrel; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: isotonic infusion
- nitrate: nitrate infusion

SUMMARY:
This study aims to investigate whether intravenous nitrate given during non-ST-elevation myocardial infarction (non-STEMI) affects the platelet inhibition of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with non-STEMI
* Patients aged 18 to 75 years
* positive troponin levels,
* blood pressure above 120/70 mmHg

Exclusion Criteria:

* Hemodynamically unstable and requiring urgent intervention,
* ST elevation on electrocardiography, atrial fibrillation,
* recurrent angina,
* use of narcotic analgesics (e.g., morphine), nitrates and glycoprotein IIb/IIIa inhibitors during hospitalization,
* history of coronary artery bypass graft (CABG) surgery,
* active infection,
* uncontrolled hypertension,
* diabetes, cerebrovascular accident, Use P2Y12 inhibitor, proton pump inhibitor, oral anticoagulant, statin, CYP enzyme-inducing or inhibiting drugs at the time of admission,
* active systemic disease (e.g., malignancy, thyroid disorders chronic inflammatory diseases, liver dysfunction),
* left ventricular systolic dysfunction (ejection fraction <50%),
* glomerular filtration rate <60 mL/min/1.73m2,
* allergy to ASA or clopidogrel, coagulopathy,
* platelet counts below 100,000/μl and hematocrit levels below 29%, or exceeding 52%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute coronary syndrome patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity Unit level | 48 hours
  Platelet Reactivity Unit <208

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Melek M, Ari H, Karakus A, Ari S, Tutuncu A, Bozat T. Impact of Intravenous Nitrate Treatment on Antiplatelet Effects of Clopidogrel in Acute Coronary Syndrome Patients: A Pilot Study. J Cardiovasc Pharmacol Ther. 2025 Jan-Dec;30:10742484251357147. doi: 10.1177/10742484251357147. Epub 2025 Jul 2. PMID 40605381